CLINICAL TRIAL: NCT01119001
Title: A P300 Brain Computer Interface Keyboard to Control Assistive Technology for People With Amyotrophic Lateral Sclerosis
Brief Title: A P300 Brain Computer Interface Keyboard to Control Assistive Technology For Use by People With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jane Huggins, PhD, Research Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H0004
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P300 Brain Computer Interface for people with ALS (Experimental)
  Interventions: Device: P300 Brain Computer Interface Keyboard

INTERVENTIONS:
Device: P300 Brain Computer Interface Keyboard — Subjects will wear an EEG cap for 1-4 hours (1-2 hours typical) per session and use the brain-computer interface to operate assistive technology. Subjects will be asked to participate in 3 sessions.
  Other Names: Electrode cap made by Electro-cap International.

SUMMARY:
People with Amyotrophic Lateral Sclerosis (ALS) will use a P300 based brain computer interface (BCI) keyboard to type in assistive technology devices. The results of this study will be compared with a previous study of a P300 BCI keyboard used by healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Diagnosed with cerebral palsy, spinal cord injury, neuromuscular disease, or ALS that results in impaired hand and arm function making it difficult to manipulate objects (if at all) and requires help to prepare or modify activities
* Able to see the BCI display
* Able to give informed consent
* Able to understand and remember instructions concerning participation
* Able to communicate effectively at least with familiar conversation partners

Exclusion Criteria:

* Are unable to give informed consent.
* Are currently experiencing open head sores
* Have a history of photo-sensitive epilepsy
* Have a history of cognitive deficits requiring accommodation or special education services
* Are unable to sit without moving the head and neck for at least 15 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Huggins, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Thompson DE, Gruis KL, Huggins JE. A plug-and-play brain-computer interface to operate commercial assistive technology. Disabil Rehabil Assist Technol. 2014 Mar;9(2):144-50. doi: 10.3109/17483107.2013.785036. Epub 2013 Apr 16. PMID 23590556

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | P300 Brain Computer Interface for People With ALS
Started | 13
Completed | 11
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | P300 Brain Computer Interface for People With ALS
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 62 [45 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Typing With a BCI Keyboard by ALS Patients.
Description: Accuracy for the sentence typed in each environment was calculated as the percentage of characters for which the result character matched the target character. The target characters were determined based on the next character needed to complete the sentence to be copied. In the case of errors, the next character was therefore a backspace to correct the error. The target characters were modified by subject comments to account for errors in selecting the next character.
  Once sentence was typed in each environment in each session on a separate day. From the three repeated sessions, there were therefore 9 total sentences per subject with 3 measures for each environment. These were treated as repeated measures for the analysis.
Time Frame: 3 times over 2-4 weeks
Measure: Mean (Full Range); unit: percentage accuracy
Groups:
- Brain-computer Interface (BCI) Environment: Accuracy typing for three sessions with the BCI acting as a stand-alone device.
- Computer Environment: Accuracy typing for three sessions with the BCI acting as a keyboard for a laptop computer.
- Assistive Technology Enironment: Accuracy typing for three sessions with the BCI acting as a keyboard for a Dynawrite communication system.
Arm/Group | Brain-computer Interface (BCI) Environment | Computer Environment | Assistive Technology Enironment
Number analyzed (Participants) | 11 | 11 | 11
percentage accuracy | 81 [41 to 100] | 78 [42 to 100] | 75 [25 to 100]

ADVERSE EVENTS:
Arm/Group | P300 Brain Computer Interface for People With ALS
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No